CLINICAL TRIAL: NCT00425425
Title: Neoadjuvant Radiochemotherapy in Local Advanced Squamous Cell Carcinoma of the Esophagus With Weekly Cetuximab Plus Oxaliplatin Plus Continuous IV. 5-FU and Conventional Fractionated External Multi-Field Irradiation up to 45 Gray. A Phase I/II Study
Brief Title: Cetuximab, Oxaliplatin, Fluorouracil, and Radiation Therapy in Treating Patients With Stage II or Stage III Esophageal Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Technical University of Munich (Other)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000516821; KRDI-TUM-OE7-432-LOR-0033-I; EU-20658; EUDRACT-2006-001097-24
Record Dates: First submitted 2007-01-19; First posted 2007-01-23 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-04

CONDITIONS: Esophageal Cancer
Keywords: squamous cell carcinoma of the esophagus; stage IIA esophageal cancer; stage IIB esophageal cancer; stage IIIA esophageal cancer; stage IIIB esophageal cancer; stage IIIC esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Squamous Cell Carcinoma | interventions — Cetuximab; Fluorouracil; Oxaliplatin; Neoadjuvant Therapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: cetuximab
Drug: fluorouracil
Drug: oxaliplatin
Procedure: conventional surgery
Procedure: neoadjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Cetuximab may also make tumor cells more sensitive to radiation therapy. Drugs used in chemotherapy, such as oxaliplatin and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving cetuximab, chemotherapy, and radiation therapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This phase I/II trial is studying the side effects and best dose of oxaliplatin and fluorouracil when given together with cetuximab and radiation therapy and to see how well they work in treating patients with stage II or stage III esophageal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of oxaliplatin and fluorouracil when administered with cetuximab and radiotherapy in patients with stage II or III squamous cell carcinoma of the esophagus. (Phase I)
* Determine the response rate in patients treated with this regimen. (Phase II)

Secondary

* Determine the toxicity of this regimen in these patients.
* Determine the postoperative complication rate and lethality in patients treated with this regimen.
* Determine the R0 resection rate in patients treated with this regimen.
* Determine the overall survival of patients treated with this regimen.
* Determine the event-free survival of patients treated with this regimen.
* Determine the metabolic response rate in patients treated with this regimen.

OUTLINE: This is a phase I, dose-escalation study of oxaliplatin and fluorouracil followed by an open-label, phase II study.

* Phase I: Patients receive cetuximab IV over 60-90 minutes on days -15, -8, 1, 8, 15, 22, and 29; oxaliplatin IV over 120 minutes on days 1, 8, 22, and 29; and fluorouracil IV continuously on days 1-5, 8-12, 15-19, 22-26, and 29-33. Patients undergo radiotherapy on days 1-5, 8-12, 15-19, 22-26, and 29-33. Patients then undergo radical esophagectomy 29-42 days after the completion of chemoradiotherapy.

Cohorts of 3-6 patients receive escalating doses of oxaliplatin and fluorouracil until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

* Phase II: Patients receive oxaliplatin and fluorouracil as in phase I at the MTD determined in phase I. Patients also receive cetuximab and undergo radiotherapy and radical esophagectomy as in phase I.

After completion of study therapy, patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 43 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous cell carcinoma of the esophagus, meeting the following criteria:

  * Locally advanced disease (T3-T4, N0-N+ [T2, N0 for cervical esophageal carcinoma])
  * Potentially resectable disease
* No distant metastases (M1b)
* No tumor infiltration of the tracheobronchial system
* Bartels preoperative risk analysis < 22

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-1 or Karnofsky PS 70-100%
* Creatinine ≤ 1.5 mg/dL OR creatinine clearance > 60 mL/min
* Bilirubin ≤ 1.5 mg/dL
* ALT and AST ≤ 2 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2 times ULN
* WBC ≥ 3,000/mm³
* Granulocyte count ≥ 2,000/mm³
* Platelet count ≥ 100,000/mm³
* No pre-existing polyneuropathy > grade 1
* No active uncontrolled infection
* PaO_2 ≥ 60 mm Hg on room air
* FEV_1 ≥ 60% of normal
* No New York Heart Association class II-IV cardiac insufficiency
* Ejection fraction ≥ 35%
* No angina pectoris (at rest or under stress) unexplained by interventional cardiology
* No myocardial infarction within the past 6 months
* No histologically confirmed liver cirrhosis
* No other malignancy within the past 5 years except carcinoma in situ of the cervix or nonmelanomatous skin cancer
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy
* No prior radiotherapy to the thorax region
* No current esophageal stent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2006-07; Primary Completion 2010-05 (Actual); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of oxaliplatin and fluorouracil (Phase I)
Response rate (histological remission) (Phase II)

SECONDARY OUTCOMES:
Toxicity as measured by NCI-CTC criteria
Postoperative complication rate and lethality
R0 resection rate
Overall survival
Event-free survival
Metabolic response rate

CONTACTS AND LOCATIONS:
Overall Officials: Florian Lordick, MD, Study Chair — Technical University of Munich
Locations (3):
- Germany (3):
  - Charite University Hospital - Campus Virchow Klinikum, Berlin
  - Universitaetsklinikum Giessen und Marburg GmbH - Marburg, Marburg
  - Klinikum Rechts Der Isar - Technische Universitaet Muenchen, Munich